CLINICAL TRIAL: NCT04446858
Title: Non-invasive Evaluation of the Predictive Value of CEUS and SWE in Patients With and Without TIPS With ACLF, Renal Failure and Hepatorenal Syndrome
Brief Title: Non-invasive Evaluation of the Predictive Value of CEUS and SWE in ACLF, Renal Failure and Hepatorenal Syndrome
Acronym: NECTAR
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Michael Praktiknjo, MD, University Hospital, Bonn
Other Study IDs: NECTAR
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Kidney Failure, Acute
Keywords: transjugular intrahepatic portosystemic shunt (TIPS); non-invasive assessments; circulating biomarkers; Transthoracic echocardiography (TTE) with Speckle-tracking; Elastography; Contrast-enhanced ultrasound; Computer tomography scan (CT-scan); Magnetic resonance imaging (MRI); Urine biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, urine, ascites, stool, DNA, PBMC, Buffi coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With TIPS: Prospective cohort that received TIPS
- Without TIPS: Prospective cohort that did not receive TIPS

SUMMARY:
Evaluation of non-invasive prognostic parameters in patients developing ACLF and renal failure in patients receiving and not receiving transjugular intrahepatic portosystemic shunt (TIPS). Patients are cared according to the local standardized follow up program. Clinical and laboratory data from standard patient care are evaluated for potential prognostic value.

DETAILED DESCRIPTION:
NECTAR consists of patients with ACLF and renal failure with and without receiving transjugular intrahepatic portosystemic shunt (TIPS) at the Department of Internal Medicine I, University of Bonn, Germany and receiving a structured routine evaluation and follow up program. The diagnosis of cirrhosis was based on clinical, hemodynamic and biochemical parameters, and ultrasound and/or biopsy criteria.

ELIGIBILITY:
Inclusion Criteria:

* All patients with portal hypertension and kidney failure

Exclusion Criteria:

* no consent, no kidney failure, no portal hypertension

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with portal hypertension and kidney failure are eligible for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Survival | up to 10 years
  death, liver transplantation

SECONDARY OUTCOMES:
Ascites | up to 10 years
  Evaluation of amount of ascites according to the Child-Score
Hepatic Encephalopathy | up to 10 years
  Evaluation of the grade according to the West Haven Criteria
Variceal Bleeding | up to 10 years
  Assessment of presence of variceal bleeding
Liver Failure | up to 10 years
  defined as Bilirubin level ≥ 12mg/dl
Acute-on-Chronic Liver Failure | up to 10 years
  Presence of ACLF according to the EASL-Chronic liver Failure Consortium (CLIF)-criteria
Kidney Failure | up to 10 years
  Assessment of AKI according to KDIGO
Organ Failures | up to 10 years
  Assessment of Organ failures according to CLIF-Sequential Organ Failure Assessment (SOFA) Score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany